CLINICAL TRIAL: NCT03780140
Title: Expanded Access to Cefiderocol for the Intravenous Treatment of Severe Gram Negative Bacterial Infections
Status: Approved for marketing | Type: Expanded Access
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Other Study IDs: S-649266-EA
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Bacterial Infections
Keywords: S-649266; cefiderocol; Gram-negative
MeSH Terms: conditions — Bacterial Infections | interventions — Cefiderocol

STUDY DESIGN:
Expanded Access Types: Individual, Intermediate

INTERVENTIONS:
Drug: Cefiderocol — Cefiderocol for intravenous infusion
  Other Names: S-649266

SUMMARY:
Expanded access may be provided for cefiderocol for qualified patients who have limited treatment options and are not eligible for a clinical trial.

ELIGIBILITY:
Hospitalized patients with serious Gram-negative bacterial infections and who have limited treatment options and are not eligible for a clinical trial.

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi

REFERENCES:
- See also: Shionogi Compassionate Use — https://www.shionogi.com/research/compassionate-use/